CLINICAL TRIAL: NCT04392687
Title: The Study of Slip Pulse Feature Extraction Method Based on the Image Processing Technology for Traditional Chinese Medicine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH107-REC2-050
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Alippery Pulse
Keywords: Wrist artery pulse diagnosis instrument; TCM pulse diagnosis; Feature extraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnoses processes of Traditional Chinese Medicine (TCM) focus on the following four main types of diagnoses methods consisting of inspection, listening and smelling, inquiry, and palpation. The most important one is palpation also called pulse diagnosis which is to measure wrist artery pulse by TCM doctor's fingers to detect patient's health state. The pulse diagnosis has three parts, namely 'Cun', 'Guan' and 'Chi', with the location. Wrist measurements correspond to different parts of the body's organs.

However, the pulse information is analyzed by TCM doctor's pulse diagnoses process, which is picked only a single waveform from a long-term pulse measured process and often discarded the other waveforms contained in the same information, e.g. Slippery Pulse waveform. The research object of this project is to divide the TCM diagnosis patients into two groups, one is the Slippery Pulse group and the other is a Normal Pulse group, in which 30 cases are collected in each group. The purpose of this project will integrate the TCM doctor's experiences and standardize them in order to construct an effective Slippery Pulse diagnosis system. It could refine Slippery Pulse diagnoses processes and reduce their diagnoses loading by using the proposed approach during this project. Therefore, we could carry out the research on feature extraction method of Slippery Pulse based on the image processing technology. We could extract the pulse characteristics of Slippery Pulse automatically from the many measurement signals and improve the automatic judging ability of the current pulse instrument to the Slippery pulse waveform. Provide important pulse information to the TCM doctors as an important reference for clinical diagnoses.

ELIGIBILITY:
Inclusion Criteria:

1. Already sign test consent permit.
2. More than 20-year-old.

Exclusion Criteria:

1. Can not accept acupuncture points stimulators.
2. Allergic to acupuncture needles.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Slippery Pulse | 30 minutes in duration.
  The purpose of this project will integrate the TCM doctor's experiences and standardize them in order to construct an effective Slippery Pulse diagnosis system.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan